CLINICAL TRIAL: NCT02179476
Title: A Multi-Site Study of the Zyga GlyDer Facet Restoration Device In Subjects With LUmbar FacET Pain Syndrome (DUET)
Brief Title: A Multi-Site Study of the Zyga GlyDer Facet Restoration Device In Subjects With LUmbar FacET Pain Syndrome - DUET
Acronym: DUET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No additional enrollment
Sponsor: Zyga Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DUET 001-003
Record Dates: First submitted 2013-01-28; First posted 2014-07-01 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Facet Joint Pain
Keywords: Facet joint; facet joint pain; facet joint disease; lumbar pain; back pain
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glyder (Experimental): Glyder Facet Restoration Device
  Interventions: Device: Glyder

INTERVENTIONS:
Device: Glyder — The Glyder Facet Restoration Device is intended for minimally invasive bilateral implantation in one or two lumbar facet levels
  Other Names: Glyder Facet Restoration Device; Glyder Device

SUMMARY:
A non-randomized, multi-site feasibility study to evaluate the safety of the Glyder Device in subjects with a history of lumbar facet joint disease (L2 to the sacrum) and successful neural ablation in which the facet joint is confirmed as the source of pain.

ELIGIBILITY:
Key Inclusion Criteria:

1. Confirmed bilateral facet joint disease demonstrated by a successful facet rhizotomy (neural ablation) within 18 months prior to enrollment
2. Facet pain is limited to one to two levels from L2 to the sacrum and pain is bilateral
3. Two diagnostic injections (MBBs) both resulting in 80% relief to confirm back pain is facetogenic
4. VAS back pain of ≥ 60 mm on a 100 mm scale, and VAS back pain is greater than or equal to the highest VAS leg pain score
5. ODI ≥ 20 points
6. At least six (6) months of non-operative conservative management (Analgesic therapy for a minimum of 2 weeks and a minimum of 4 weeks of NSAID therapy; Supervised exercise and/or physical therapy program-minimum of 12 sessions)
7. At least 22 years of age and skeletally mature

Key Exclusion Criteria:

1. Pain is from a spinal structure other than facet joints (i.e., disc, hip and SI joint pain are excluded)
2. Osteoporosis or severe osteopenia
3. Lumbar fusion
4. Symptomatic spinal stenosis requiring surgical intervention
5. Prior total disc replacement, fusion, decompressive laminectomy, facetectomy, or placement of a posterior spinous process device
6. Disc herniation requiring surgical intervention
7. The subject has a Body Mass Index (BMI) of greater than 35
8. Planned elective surgery within 12 months

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-06; Primary Completion 2017-12 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 6 months
  Safety will be evaluated by assessing the incidence of device and/or procedure related serious adverse events.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - The Spine Institute, Santa Monica, California
  - Laser Spine Institute, Tampa, Florida
  - Clinical Radiology of Oklahoma, Edmond, Oklahoma
  - Northwest Orthopaedic Specialists, Spokane, Washington